CLINICAL TRIAL: NCT01818037
Title: A Long-term Postoperative Outcome After Bilateral Congenital Cataract Surgery in Eyes With Microphthalmos
Brief Title: Long-term Postoperative Outcomes After Bilateral Congenital Cataract Surgery in Eyes With Microphthalmos
Status: Completed | Type: Observational
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, Director, Iladevi Cataract and IOL Research Center, Iladevi Cataract and IOL Research Center
Other Study IDs: 13-002
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Microphthalmos With Congenital Cataracts
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Microphthalmos with congenital cataract: 72 eyes of 36 patients with microphthalmos who underwent bilateral congenital cataract surgery between January 2003 and June 2008.
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery

SUMMARY:
Cataract surgery in infantile eyes, which are microphthalmic, can be even more demanding.

In addition, the frequent presence of other ocular and systemic anomalies such as nystagmus, glaucoma, amblyopia, and higher rate of postoperative complications may limit the success of cataract surgery.

In our previous study, the investigators examined the intraoperative performance and postoperative outcomes of bilateral cataract surgery in microphthalmic eyes of patients before their first birthday. At 1 year, the postoperative results showed that good visual outcomes could be obtained in microphthalmic eyes.

Since only a few studies have reported outcomes, and that too only short term of cataract surgery on microphthalmic eyes, in this prospective observational study we evaluated the long-term impact of bilateral cataract surgery on eyes with microphthalmos. The investigators examined the outcomes, complication rates, influence of age at surgery on pattern of axial growth and central corneal thickness and visual and orthoptic assessment in these eyes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of microphthalmos and congenital cataract.
* Microphthalmos was defined as an eye with an axial length (AL) that is more than 2 SD smaller than the normal for that age group according to Gordon and Donzes

Exclusion Criteria:

- Children with congenital anomalies such as posterior persistent fetal vasculature causing stretching of the ciliary processes or a tractional retinal detachment, aniridia, and chorioretinal coloboma were excluded.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 72 eyes of 36 patients with microphthalmos who underwent bilateral congenital cataract surgery between January 2003 and June 2008.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2003-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Glaucoma following cataract surgery | 45 months postoperative

SECONDARY OUTCOMES:
Posterior synechiae | 45 months postoperatively
visual axis obscuration | 45 months
axial length rate of growth | 45 months postoperatively
central corneal thickness | 45 months postoperatively
visual acuity | 45 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Iladevi Cataract & IOL Research Center, Ahmedabad, Gujarat, India